CLINICAL TRIAL: NCT06877598
Title: Canada-wide Implementation of a Virtual Sexual Health and Rehabilitation eClinic (SHAReClinic) for Prostate Cancer Patients and Their Partners
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 708251
Record Dates: First submitted 2025-03-06; First posted 2025-03-14 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Sexual Dysfunction, Physiological; Sexual Dysfunction, Psychological; Sexual Dysfunction; Virtual Care; Virtual Clinic; Survivorship; Implementation of Evidence Based Programs; Implementation
Keywords: Sexual Dysfunction; Prostate cancer; Virtual health; Implementation; Consolidated Framework for Implementation Research (CFIR); Bio-psychosocial; Reach Effectiveness Adoption Implementation and Maintenance (RE-AIM); Survivorship
MeSH Terms: conditions — Prostatic Neoplasms; Sexual Dysfunction, Physiological; Sexual Dysfunctions, Psychological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate the effectiveness of SHAReClinic, a national, virtual Sexual Health and Rehabilitation eClinic designed to support prostate cancer patients and their partners. Specifically, this study aims to assess SHAReClinic's impact on improving sexual function, satisfaction, and relational intimacy after treatment.

The primary objective is to evaluate SHAReClinic's effectiveness across participating sites and determine its role in supporting long-term sexual health and well-being.

As part of usual care, newly enrolled SHAReClinic patients will receive guided education modules and access to sexual health counselling at key recovery milestones.

SHAReClinic seeks to expand access to sexual health care for prostate cancer patients across Canada by providing evidence-based, virtual sexual rehabilitation. Findings from this study will inform best practices in survivorship care and contribute to the development of a national standard for oncology sexual health interventions.

DETAILED DESCRIPTION:
Detailed Description The considerable prevalence of sexual dysfunction (SD) after prostate cancer (PCa) treatment makes SD post-treatment a substantial health-related quality of life burden for patients and their partners. Research indicates that 40% to 75% of men suffer from SD post-PCa. Sixty percent of men experience significant distress in response to SD. Significant distress is also reported by partners and couples. Overall, patients cite sexual health concerns as the most significant unmet need following treatment for PCa. Accordingly, there is an existent need for equitable, timely, and affordable access to high-quality SD treatment for Canadian PCa patients and their partners.

Unfortunately, none of the empirically-based, comprehensive interventions reported in the literature have been implemented into clinical settings in Canada. The lack of translation from research evidence to clinical implementation is common across healthcare provision. It is known that most research, even positive full-scale studies, do not result in practice-change or take years to do so. A key aspect contributing to this lack of knowledge translation is the complexity of transitioning an "experimental intervention" to "real world" clinical settings. In sexual healthcare in oncology, ineffective knowledge translation is ubiquitous and includes several unique complexities that impair the implementation, integration, and sustainability of empirically-based treatment.

The recent advent of virtual care in healthcare offers an opportunity to address many of the barriers to implementing sexual recovery programs within PCa treatment facilities. Virtual care provides greater accessibility for patients not proximal to cancer centres, or who are unable to travel due to financial constraints or physical limitations. Encouragingly, examples of internet-delivered interventions exist for men with PCa and their partners. Schover and colleagues found that a digitally-based intimacy enhancement intervention was as effective as a brief in-person sex therapy intervention in improving sexual outcomes in couples after PCa. Although these advances in models of care provision are inspiring, the majority of Canadian PCa patients and their partners have yet to benefit from virtual care innovations.

In an effort to advance evidence-based survivorship programming in the treatment of SD post-PC, a team of expert Canadian healthcare practitioners and patient/partner advocates developed the Sexual Health and Rehabilitation eClinic (SHAReClinic). SHAReClinic is a web-based, bio-psychosocial SD intervention specifically for patients/couples who have undergone treatment for PCa. A pilot study evaluating the acceptability and engagement of SHAReClinic achieved significant patient activity on the platform and 80% patient engagement at 1-year follow-up. Additionally, evaluation of the effectiveness of SHAReClinic showed non-inferior sexual health outcomes when compared to a "best practice" in-person sexual health clinic.

Rationale Sexual dysfunction after PCa treatment has significant adverse impacts on patient/partner health-related quality of life. Few Cancer Centres in Canada offer comprehensive care for SD post-PCa treatment, resulting in significant barriers to care equity and access. SHAReClinic is established as effective virtual care programming for SD post-PCa.

The goal of this research is to evaluate the SHAReClinic in 2 cancer centres currently using it as usual care and 9 cancer centres which has newly implemented SHAReClinic as part of their usual care. The SHAReClinic will be offered to 1. Newly diagnosed patients at who are scheduled to undergo active treatment for localized prostate cancer, 2. patients currently undergoing active treatment for prostate cancer and 3. patients who have undergone prostate cancer treatment within the last 6 months. Active treatment can include any of the following options surgical, radiation, and/or ADT. The SHAReClinic goals are to re-establish optimal sexual function, satisfaction and to support the maintenance of intimacy following prostate cancer treatment. These goals are addressed through two complementary components: 1) a bio-medical component (erectile rehabilitation), focused on the long term penile health or short-term erectile function as per patient preference, and 2) a psychological component (intimacy maintenance), involving the maintenance or restoration of couples' intimacy and sexual activity (penetrative or non-penetrative). Both physical and psychological factors can affect patients' sexual satisfaction after cancer treatment; resultantly, interventions should incorporate a bio-psychosocial approach to rehabilitation.

Study Design This is a prospective observational evaluation of a virtual sexual health and rehabilitation intervention program. As part of patient standard care, facilitated web-based clinic visits will be provided to patients once before treatment, 6 weeks, 10 weeks, 4 months, 6 months and 12 months post cancer treatment. Patients who opt-in to the SHAReClinic will also be invited to register for this study. The study involves no additional requirements from patients, as all questionnaires (baseline, 6-weeks, 6 months, and 12 months) are completed as part of their enrolment in the SHAReClinic.

Patients experience in the SHAReClinic involves the following: Upon registration, patients will be paired with a sexual health coach from their center and asked about their availability to receive a phone/video call from their sexual health coach. At the beginning of the first clinic visit, participants will be asked to complete a set of questionnaires. The questionnaires take around 10-15 minutes to complete. Patients are also asked to complete the same questionnaires at 6 week, 6 months and 12 months. The topics covered in each clinic visit vary and are based on the treatment schedules of the participants. A Q&A session on the web page will be available for participants to leave any questions or concerns regarding their sexual health, rehabilitation process and the content of the portal. Participants are free to request for a check-in call with their sexual health coach if they want to chat about their concerns by phone. Each clinic visit will last approximately 30 minutes. If participants miss their clinic visit, they will get a notification from the platform and then a reminder call from their sexual health coach. At the end of their final SHAReClinic clinic visit, participants will be asked to fill out a satisfaction questionnaire, including questions about the ease of access to the website, their experience with SHAReClinic portals and communication with their sexual health coach. The satisfaction questionnaire takes about 10 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for first-line treatment for localized prostate cancer, either through radical prostatectomy (open or robotic) or radiation treatment (brachytherapy, external beam) Alone, or with adjuvant Androgen Deprivation Therapy (ADT) OR

  * Patients currently undergoing active treatment for prostate cancer OR
  * Patients who have undergone cancer treatment in the past 6 months
  * Patients who are hormone and/or chemotherapy-naïve
  * Patients who have access to a computer or smartphone with internet access
  * Patients who are 18 years of age or older

Exclusion Criteria:

* Patients on ADT alone as primary treatment, and/or patients on chemotherapy
* Patients who lack English proficiency
* Patients on nitrate therapy or have other contra-indications to phosphodiesterase type 5 inhibitors (PDE5i's)
* Patients with medical conditions that would preclude safe sexual activity
* Patients who have had previous treatment for PCa

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of newly enrolled SHAReClinic patients across the 11 participating cancer centers. These participants will be prostate cancer patients who are either about to start, currently undergoing, or have recently completed treatment. The study will assess their experiences and outcomes as they engage with SHAReClinic as part of their usual care.
Sampling Method: Non-Probability Sample
Enrollment: 575 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Assessing SHAReClinic's Impact on Sexual Function and Satisfaction | Baseline, 6 weeks, 6 months, and 12 months
  Measured using: PROMIS-20 Full Profile Sexual Function and Satisfaction (Male)
  This outcome assesses sexual function and satisfaction across multiple domains, including erectile function, orgasm, and overall sexual activity. Each item is scored on a 5-point Likert scale, and raw scores are converted to T-scores (Mean = 50, SD = 10). A higher T-score indicates better sexual function and satisfaction. The measure is collected at multiple time points to track changes in sexual function over time.
Assessing SHAReClinic's Impact on Sexual Distress | Baseline, 6 weeks, 6 months, and 12 months
  Measured using: Sexual Distress Scale (SDS - Male)
  This outcome measures the level of distress related to sexual function, including anxiety and emotional responses to changes in sexual activity post-treatment. Items are rated on a 5-point scale, and total scores are summed. A higher score indicates greater sexual distress, meaning that patients experiencing more distress will have higher numerical values. This outcome is assessed periodically to evaluate changes over time.
Assessing SHAReClinic's Impact on Relational Intimacy | Baseline, 6 weeks, 6 months, and 12 months
  Measured using: Miller Social Intimacy Scale (MSIS)
  This outcome evaluates emotional and physical intimacy between partners. The scale measures the frequency and intensity of intimate interactions, providing insight into relationship closeness post-treatment. Items are rated on a 10-point scale, with total scores summed to create an overall intimacy score. Higher scores indicate greater relational intimacy. This measure helps determine how SHAReClinic interventions impact the intimacy of participants and their partners.
Assessing SHAReClinic's Impact on Health-Related Quality of Life | Baseline, 6 weeks, 6 months, and 12 months
  Measured using: Expanded Prostate Index Composite Short Form (EPIC-26)
  This outcome assesses multiple domains of health-related quality of life, including urinary, bowel, sexual, and hormonal function. Scores for each domain are transformed linearly to a 0-100 scale, where higher scores indicate better quality of life in that domain. The EPIC-26 allows for a comprehensive evaluation of how SHAReClinic impacts sexual health and broader survivorship concerns.
Overall Patient Satisfaction with SHAReClinic | Final clinic visit (12 months)
  Measured using: SHAReClinic Satisfaction Questionnaire
  This outcome measures participant satisfaction with the SHAReClinic platform and its interventions. Patients rate their satisfaction with various aspects of the program, including ease of access, quality of resources, and effectiveness of support services. Items are scored on a 5-point Likert scale, where higher scores indicate greater satisfaction. This measure is collected at the end of the study to assess the overall user experience.

SECONDARY OUTCOMES:
System-Level Evaluation: Enrolment, Attrition, and Adherence Rates | From enrollment to the end of 1st year on SHAReClinic
  This objective evaluates the feasibility and sustainability of SHAReClinic by analyzing recruitment, retention, and adherence trends.
  How This Is Measured:
  Enrolment rates → Number of patients registering for SHAReClinic at each site. Attrition rates → Number of patients who discontinue SHAReClinic participation before completing the full program.
  Adherence rates → Number of patients who complete all scheduled clinic visits (6 total) within the 12-month follow-up.
Evaluating Patient Interest and Acceptance of SHAReClinic | From enrollment to the end of 1st year on SHAReClinic
  SHAReClinic's success depends on its acceptability and usability among prostate cancer survivors.
  How This Is Measured:
  Recruitment Interest → Tracked by number of patients who register for SHAReClinic upon referral.
  Patient Acceptance (Attrition Analysis) → Measured through dropout rates, patient-reported reasons for withdrawal, and qualitative feedback.
Data Completeness and Quality | From enrollment to the end of 1st year on SHAReClinic
  Ensuring that all patient-reported data is collected and available for analysis.
  How This Is Measured:
  Clinic visit completeness → Percentage of patients who complete six months/one year clinic visits.
  Data completeness → Percentage of patients who submit all required PROMIS SexFS, EPIC-26, SDS, and MSIS questionnaires.
  Integrity of data collection → Tracked by missing or incomplete responses. Comparison of data consistency across sites → Evaluates whether data is collected uniformly across all 11 cancer centers.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Matthew, PhD. C.Psych, Principal Investigator — Princess Margaret Cancer Centre
Locations (10):
- Canada (10):
  - Vancouver Coastal Health Authority, Vancouver, British Columbia
  - Men's Health Clinic Manitoba, Winnipeg, Manitoba
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Dianne & Irving Kipnes Urology Centre, Edmonton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - St. Joseph's Health Care London, London, Ontario
  - Trillium Health Partners, Mississauga, Ontario
  - Grass Family Men's Health Center, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - St. Paul's Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No